CLINICAL TRIAL: NCT05775874
Title: A Sigle-arm，Open Label，Multicenter Study of AZD4547 Combination With Tislelizumab for Patients With Metastatic or Locally Advanced Urothelial Carcinoma (mUC) Harboring Fibroblast Growth Factor Receptor Alterations
Brief Title: A Study to Evaluate the Safety and Efficacy of AZD4547 Combination With Tislelizumab in Patients With mUC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK091-203
Record Dates: First submitted 2022-10-08; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — AZD4547; tislelizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- An open evaluation of AZD4547 combined with Tislelizumab in UC patients (Other): AZD4547 : Initiation dose 80mg BID,po;Until disease progression, death, loss to follow-up, voluntary withdrawal of informed consent, development of intolerable toxicity, investigator decision to discontinue treatment, or completion of the entire study.
  Tislelizumab:200mg Q3W, Until disease progression, death, loss to follow-up, voluntary withdrawal of informed consent, development of intolerable toxicity, investigator decision to discontinue treatment, or completion of the entire study.
  Interventions: Drug: AZD4547; Drug: Tislelizumab

INTERVENTIONS:
Drug: AZD4547 — Initiation dose: 80mg BID,po.
  Other Names: FGFR1/2/3/4 inhibitor
Drug: Tislelizumab — Tislelizumab:200mg Q3W
  Other Names: PD1 inhibitor

SUMMARY:
This trial is an open, phase II clinical study. The study is divided into two parts: A and B, and the part A evaluate the safety and tolerability of AZD4547 combined with Tislelizumab in patients with locally advanced or metastatic urothelial cancer, determine the recommended dose of midoral AZD4547 combined with Tislelizumab in a Chinese patient population. Part B study will evaluate the efficacy of this recommended dose combined with Tislelizumab in patients with locally advanced or metastatic urothelial cancer with FGFR2 / 3 alterations , and will also further evaluate the safety, tolerability, and PK and PD characteristics of AZD4547 in combination with Tislelizumab.

DETAILED DESCRIPTION:
Part A of the study In Part A, subjects will receive AZD4547 80mg BID orally for cycles every 21 days and terelizumab 200mg will be an intravenous infusion (IV) 200mg every 3 weeks. Subsequent subjects in Part A should be administered at least 7 days after the first dose of the first subject (sentinel subject). . Tolerability will be assessed based on the incidence of dose-limiting toxicity (DLT) observed in cycle 1 (21 days). Part B; If a DLT event occurs in> 1 of the 6 DLT-evaluable subjects, With the consent of the investigator and the sponsor, An additional combined regimen cohort of six patients with a lower AZD4547 dose (AZD4547 60mg BID + Tislelizumab 200mg Q3W) will be initiated. I A specific dose / regimen of subjects and no more than one subject with DLT events will be selected to confirmation for confirmation for use in the Part B study. After cycle 1, subjects will continue to receive combination therapy in one cycle every 21 days until disease progression, death, loss to follow-up, voluntary withdrawal of informed consent, occurrence of intolerable toxicity, investigator decision to terminate treatment, or the end of the entire study. Safety assessments will be performed in each visit cycle, including the incidence and severity of adverse events (according to CTCAEv5.0) and laboratory abnormalities Study Part B Patients with locally advanced or metastatic urothelial carcinoma harboring FGFR2 / 3 alterations will follow the Simon's optimal two-stage design. It was considered "efficacy evaluable" when tumor assessment results were available at both baseline and after treatment

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this clinical trial, understand the study procedures, and be able to sign a written informed consent.
2. Age of 25 years old at the time of signing the informed consent (or the age range specifically required by the regulatory agency or ethics), without gender limitation;
3. By histologically confirmed, surgical unresectable local advanced or metastatic urothelial cancer patients, can be accompanied by other histological type differentiation (including adenoid, squamous or other types)
4. The ECOG PS (performance status) score is 0-1 point;
5. The estimated survival period of 3 months;
6. Good organ function level meets the following laboratory examination requirements, and the examination results should be obtained within 14 days before the first administration of the study treatment
7. Fertility female or male subjects must agree to use a medically approved contraceptive measure during the study treatment and within 6 months after the end of the study treatment period; fertile female subjects must have a negative blood β -hCG test within 7 days before the first dose and must be non-lactating;

Exclusion Criteria:

1. Known allergic to AZD4547 tablets or components; allergic to monoclonal antibody drugs and fusion protein drugs.
2. Patients with imaging progression after previously receiving selective FGFR inhibitors or receiving immune checkpoint inhibitors
3. Subjects with a history of an active autoimmune disease or a possible recurrence of an autoimmune disease, as judged by the investigator, should be excluded. Patients are admitted for the following diseases: hypothyroidism that can be controlled by hormone replacement therapy only, skin diseases without systemic treatment
4. A history of idiopathic pulmonary fibrosis (including pneumonia), drug-related pneumonia, organic pneumonia
5. Subjects requiring systemic treatment with corticosteroids (prednisone or similar drug> 10 mg / day) or other immunosuppressive agents within 14 days prior to enrollment.a)
6. Other malignant tumors requiring treatment were present within 6. 3 years

7 The electrolyte disorders that cannot be corrected and affect serum potassium, blood calcium or blood phosphorus levels.

8. Unstable or symptomatic CNS transfer

9. The researchers judge that the subject has factors that significantly affect the absorption of oral drugs.

10 Current active infection or fever of unknown origin> 38.5℃

11. Previous allograft or stem cell transplantation or organ transplantation.

12. Use of any live or attenuated vaccine against infectious diseases (e. g., influenza, chickenpox, etc.)

13. End time of other anti-tumor treatment from first study drug:

14. Patients with reversible adverse events caused by previous antitumor therapy, not returning to grade CTCAE

15 Patients are using, or are using, the following drugs or foods within 7 days before the first administration of the study treatment: CYP3A4 and CYP2D6 strong inhibitors or inducers.

16. Presence of uncontrolled cardiovascular disease or medical history, including: a) Congestive heart failure

17. Any abnormal corneal or retinal changes that may increase the risk of ocular toxicity during screening, including:

18. Human immunodeficiency virus (HIV) infection (HIV antibody serotest positive) or previously acquired / hereditary immunodeficiency disease

19 Patients with refractory / uncontrolled ascites or pleural effusion. Patients were allowed to use an indwelling catheter.

20 Severe unhealed skin / mucosal ulcers, chronic ulcers of the lower extremities, known gastric ulcers, or incisions are present.

21. Any other medical treatment (e. g., respiratory, metabolic, infectious, immune, congenital, endocrine, or central nervous system diseases), mental or social factors that may sign informed consent, cooperation, participate in clinical studies or affect the interpretation of the research results.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety index | At the end of Cycle 1 (each cycle is 28 days)
  Part A:Dose limiting toxicity (DLT) incidence
Effectiveness indicators | at least 8 weeks
  Part B: Objective remission rate

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China